CLINICAL TRIAL: NCT01645254
Title: Phase 1b Clinical Trial Using Argemone Mexicana in Healthy Adults Infected or Not Infected With Plasmodium Falciparum in Mali: Pharmacokinetics and Observational Study
Brief Title: Phase 1b Malaria Clinical Trial Using Argemone Mexicana in Healthy Adults in Mali
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Bamako (Other)
Collaborators: University of Geneva, Switzerland (Other)
Responsible Party: Principal Investigator, Issaka Sagara, M.D., MSPH, Principal Investigator, University of Bamako
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MRTC_Arge01; MRTC_Arge01 (Other: MRTC_Arge01)
Record Dates: First submitted 2012-07-03; First posted 2012-07-20 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Malaria
Keywords: healthy volunteers; pharmacokinetics; malaria; Argemone mexicana
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Argemone mexicana (Experimental): Argemone mexicana is traditional medicinal plant known as having an antimalarial activity.
  The aerial part of this plant is used. The decoction of the powder of the plant will be used.
  Interventions: Drug: Argemone mexicana

INTERVENTIONS:
Drug: Argemone mexicana — 30g, the powder decoction 2 times a day for 14 days
  Other Names: traditional antimalarial

SUMMARY:
The main objective is to study the pharmacokinetics, pharmacodynamics and tolerability of the decoction of the aerial parts of Argemone mexicana (AM), administered in healthy volunteers.

DETAILED DESCRIPTION:
This is an open non comparative safety and pharmacokinetic (PK) study clinical trial. Healthy volunteers aged from 18 to 50 years old will be recruited and followed 42 days after treatment initiation as in the current World Health Organization malaria drug protocol efficacy assessment protocol.

Each volunteer will be take oral Argemone mexicana in decoction formulation. For the PK assessment purposes, 3 groups have been constituted: (i) a group will receive a unique dose of with blood withdrawal scheduled at 0 hour, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hour , 8 hours and 12 hours. (ii) a group will receive two doses (morning and evening) of Argemone mexicana for 14 days with blood withdrawal scheduled at 0 hours, 30 minutes, 1 hour, 2 hours, 4 hours, 6 hours, 8 hours, 12 hours, 24 hours, 3 days, 7 days and 14 days. (iii) a group will receive two doses (morning and evening) of Argemone mexicana for 14 days with blood withdrawal scheduled at 0 hour, 12 hours, 14 hours, 16 hours, 18 hours, 20 hours, 22 hours, 24 hours, 3 days, 7 days, 14 days and 21 days Safety will be assessed clinically (Clinical exam and Electrocardiography) and biologically (hematology and biochemistry parameters will be measured) throughout the 42 days of thefollow-up.

ELIGIBILITY:
Inclusion Criteria:

* age of 18-50 years old;
* be in good general health;
* be available for the duration of the study;
* agreement to participate in the study
* be a resident of the village known study;
* acceptance of the conservation laboratory specimens for future research.

Exclusion Criteria:

* Plasmodium falciparum infection with clinical manifestations;
* Presence of severe or complicated malaria;
* Acute medical condition;
* Any other medical condition that requires medical attention inconsistent with the study or interfere with the study;
* Severe medical conditions;
* Allergy to the product of the study,
* Pregnant women or nursing
* Taking a derivative product of the study or other known antimalarial within 14 days before enrollment.
* Refusal to participate

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-09; Primary Completion 2012-10 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Number of Adverse Events | 6 weeks
  health volunteers will be assessed daily for 3 days and then on Day 7 and then weekly up to 6 weeks.

SECONDARY OUTCOMES:
Plasma concentration curves of the drug | 6 weeks
  The phramacokinetics measured will be performed depending on the treatment groups. Three different treatment groups have constituted, each group will be allocated a specific time point for PK assessment.

CONTACTS AND LOCATIONS:
Overall Officials: Issaka Sagara, MD,MSPH, Principal Investigator — University of Bamako
Locations (1):
- Malaria Research and Training Center, USTTB, Bamako, Mali